CLINICAL TRIAL: NCT03189979
Title: Club Fit: Pilot Testing of a Physical Activity and Healthy Eating Intervention at a Boys & Girls Club After School Program
Brief Title: Club Fit: Physical Activity and Healthy Eating at an After School Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Mark L Wieland, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-003639; UL1TR000135 (NIH)
Record Dates: First submitted 2017-06-15; First posted 2017-06-16 (Actual); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Childhood Obesity; Physical Activity; Dietary Habits
Keywords: community based participatory research; Childhood obesity
MeSH Terms: conditions — Pediatric Obesity; Motor Activity; Feeding Behavior | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Club Fit (Experimental): Intervention includes exposure to physical activity and healthy eating intervention policy implementation, staff training, a challenge/self-monitoring program for healthy behaviors, a peer-coaching program for healthy behaviors, and a social marketing campaign.
  Interventions: Behavioral: Physical activity and healthy eating intervention

INTERVENTIONS:
Behavioral: Physical activity and healthy eating intervention — Using a community-based participatory approach, BGC staff and academic researchers developed intervention components informed by formative studies and based on a social ecological theory framework. Components included healthy eating and physical activity policy implementation, staff training, a challenge/self-monitoring program for healthy behaviors, a peer-coaching program for healthy behaviors, and a social marketing campaign.
  Other Names: Club Fit

SUMMARY:
Background: Youth from low-income and minority families are disproportionately affected by obesity and its complications. This study presented pilot work to develop and implement a multi-component physical activity and healthy eating intervention at a Boys & Girls Club (BGC) after school program.

Methods: Using a community-based participatory approach, BGC staff and academic researchers developed intervention components informed by formative studies and based on a social ecological theory framework. Components included healthy eating and physical activity policy implementation, staff training, a challenge/self-monitoring program for healthy behaviors, a peer-coaching program for healthy behaviors, and a social marketing campaign. Preliminary intervention efficacy was assessed through a single group, pre-post study design with measured collected at baseline and 6 months.

ELIGIBILITY:
Inclusion Criteria:

- Active Boys & Girls Club participation, which was defined as expected Club attendance at least twice weekly.

Exclusion Criteria:

- None

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 61 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Change in self-efficacy | baseline, 6 months
  Self-efficacy was assessed with a survey adapted from instruments developed for the Patient-centered Assessment and Counseling for Exercise plus Nutrition program for low-income, ethnically diverse adolescents. It was scored on a 10-point Likert scale from 1 (not at all confident) to 10 (extremely confident).
Change in motivation | baseline, 6 months
  Motivation for physical activity was scored on a 10-point Likert scale from 1 (not at all motivated) to 10 (extremely motivated).

SECONDARY OUTCOMES:
Change in body mass index | baseline, 6 months
  For body mass index (BMI), weight was measured to the nearest 0.1 kg using a single scale. Height was measured to the nearest 0.1 cm using a stadiometer. BMI was calculated as weight (kg)/height squared (m2).
Change in physical activity | baseline, 6 months
  The Kinetic Activity Monitor accelerometer was used for objective physical activity assessment. Participants were asked to wear the accelerometer at their waist during waking hours for 10 consecutive days. The accelerometer was activated and data collected without providing feedback to participants. A valid assessment required 5 days of wear for at least 10 hours a day. Data output included sedentary time and time spent performing mild, moderate, and vigorous physical activities.
Change in dietary quality | baseline, 6 months
  Dietary assessment was performed with the Beverage and Snack Questionnaire 2. The instrument was adapted to include nine items (on a 7-point Likert scale) that addressed consumption of fruits, vegetables, and sugar sweetened beverages. The Likert scale ranged from "never or less than 1 per week" to "4+ per day." The greater number of fruits and vegetables, and fewer number of sugar sweetened beverages were considered a positive change in dietary quality.

CONTACTS AND LOCATIONS:
Overall Officials: Mark L Wieland, MD, MPH, Principal Investigator — Mayo Clinic
Locations (1):
- Boys & Girls Club of Rochester, MN, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared.